CLINICAL TRIAL: NCT05382767
Title: A Randomized, Double-blind, Active-controlled, Multicenter Phase I Trial to Investigate the Safety and Efficacy of CKDB-501A in Subjects With Post-stroke Upper Limb
Brief Title: Safety and Efficacy of CKDB-501A in Subjects With Post-stroke Upper Limb Spasticity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CKD Bio Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CKDB-BAUL-101
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Post-stroke Upper Limb Spasticity
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CKDB-501A (Experimental)
  Interventions: Drug: CKDB-501A
- Botox® (Active Comparator)
  Interventions: Drug: Botox®

INTERVENTIONS:
Drug: CKDB-501A — Muscle Spasticity
  Arms: CKDB-501A
Drug: Botox® — Muscle Spasticity
  Arms: Botox®

SUMMARY:
Multicenter, randomized, double-blind, active-controlled, parallel-design study to evaluate the safety and efficacy of CKDB-501A in Subjects with Post-stroke Upper Limb Spasticity

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 19 years
* History of stroke more than 24 weeks prior to screening
* ≥ 2 points in the focal spasticity of wrist flexor and ≥ 1 point at least one of finger flexor and elbow flexor as measured on MAS(0 to 4)
* ≥ 2 points in one of the targeted functional disability item (i.e. hand hygiene, clothing, upper extremity, or pain for evaluation on DAS

Exclusion Criteria:

* Neuromuscular disorders such as Lambert-Eaton syndrome, myasthenia gravis, or amyotrophic lateral sclerosis
* Fixed joint/muscle contracture in the target limb
* History(within 24 weeks of screening visit) or planned(during study period) treatment with phenol or alcohol injection(chemodenervation) or surgery in the target limb
* History(within 4 months of screening visit) or planned(during study period) treatment with tendon lengthening in the target limb
* History(within 12 weeks of screening visit) treatment with Botulinum Toxin
* Concurrent treatment with an intrathecal baclofen
* Known allergy or sensitivity to the study medication or its components (Clostridium botulinum toxin type A, albumin, Sodium chloride, etc.)
* Male and Female who are not willing to take any appropriate means of contraception during the study period
* Patients who are not eligible for this study at the discretion of the investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | up to week 12
  severity and frequency of reported adverse events

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No